CLINICAL TRIAL: NCT07248878
Title: Pilot Study for the Generation of Cervical Cancer Organoids From Patients Undergoing Diagnostic Biopsy
Acronym: Cervical organ
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Università di Verona, AOUI Verona Dipartimento di Ostetricia e Ginecologia (Unknown)
Responsible Party: Sponsor
Other Study IDs: RS315/IRE/25
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Stage IB2; Cervical Cancer Stage IIa; Cervical Cancer Stage IB; Cervical Cancer Stage IIIA
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, tissue sample, vaginal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected cervical cancer: Patients with a suspected diagnosis of cervical cancer for whom a biopsy is indicated according to clinical practice who undergo a biopsy at the Gynecological Oncology Unit of the Regina Elena Cancer Institute in Rome.

SUMMARY:
A meta-analysis showed that neoadjuvant chemotherapy followed by radical hysterectomy reduces the risk of mortality by 35% compared to radiotherapy alone, with a 14% increase in five-year survival. Unfortunately, however, approximately 30% of patients undergoing neoadjuvant chemotherapy are referred for adjuvant radiotherapy or chemoradiotherapy due to the presence of high recurrence risk factors after surgery, which results in a bi- or tri-modal treatment with very serious consequences in terms of toxicity. Infact, approximately 20% of patients treated with radiotherapy experience vaginal discomfort up to 3 years after completing treatment, with significant consequences for the women's quality of life. Therefore, on the one hand, it would be appropriate to identify new drugs that synergize with chemotherapy, reducing the need for adjuvant radiation; on the other, it could be useful to identify patients who could truly benefit from neoadjuvant treatment. To do this, it is necessary to have ex vivo biological models capable of simulating the complexity of the tumor environment and that can be used as a tool to investigate tumor response to specific treatments.

In this context, tumor organoids represent ideal alternative in vitro models, capable of preserving the characteristics of the original tumors, including their architecture and cell types present. They can be used as avatars for the selection of specific anticancer therapies and for the creation of patient biobanks.

DETAILED DESCRIPTION:
The study involves the prospective recruitment of patients with suspected cervical cancer who undergo a biopsy at the Gynecological Oncology Unit of the Regina Elena Cancer Institute in Rome. Patients will be given an explanation, reading, and signing of the informed consent form.

They will undergo a biopsy and tissue sampling according to clinical practice during colposcopy.

A vaginal swab and blood sample will be taken before the biopsy. The tissue collected during the biopsy will be analyzed, and cases of cervical cancer with FIGO IB2, IB3-IIA2, and IIA1 or FIGO III will be selected for organoid culture.

If the analyzed tissue is negative for the presence of cancer (approximately 2% of cases), the patient will be considered a screening failure.

A portion of the tissue (approximately 1 cm) and the collected blood, only if their availability and adequacy are guaranteed for the purpose of conserving suitable material in an archive, will be sent to the IRE Translational Oncology Research Laboratories and used for the generation of organoids. The vaginal swab will be sent to the ISG Microbiology and Virology Laboratory for microbiome analysis.

The blood, tissue, and swab collected for patients who fail to respond will remain available to the IRE Anatomy Pathology Unit or will be biobanked for future studies related to this project.

ELIGIBILITY:
Inclusion Criteria:

* female over 18 years of age;
* suspected diagnosis of cervical cancer for which a biopsy is indicated according to standard clinical practice;
* Informed consent (study participation and data processing) given in writing personally and/or through the legal representative/guardian/support administrator/witness, before any study-specific procedure is performed.

Exclusion Criteria:

* previous malignancies;
* previous systemic treatments;
* previous antibiotic treatment before surgery. Any antibiotic treatment must be stopped at least 3 weeks before surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with a suspected diagnosis of cervical cancer for whom a biopsy is indicated
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
RNA-sequencing | 36 months
  DNA for WES profiling will be extracted from biopsy tissue and PDOs using the AllPrep kit.
  The DNA/RNA/miRNA Universal Kit will be used to prepare organoid cultures.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided